CLINICAL TRIAL: NCT04766333
Title: NJ HEROES TOO (New Jersey Healthcare Essential Worker Outreach and Education Study - Testing Overlooked Occupations)
Brief Title: New Jersey Healthcare Essential Worker Outreach and Education Study - Testing Overlooked Occupations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Shawna V. Hudson, PhD, Professor and Research Division Chief Department of Family Medicine and Community Health, Rutgers, The State University of New Jersey
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2020002549; 3UL1TR003017-02S2 (NIH)
Record Dates: First submitted 2021-02-10; First posted 2021-02-23 (Actual); Results first posted 2023-03-10 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Covid19; Health Care Seeking Behavior; Health Behavior
MeSH Terms: conditions — COVID-19; Patient Acceptance of Health Care; Health Behavior

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthcare Worker Focused Outreach Intervention Strategy (Active Comparator): Healthcare Worker Focused Outreach Intervention Strategy
  Interventions: Behavioral: Healthcare Worker Focused Outreach
- Community Organization Led Outreach (Active Comparator): Community Organization Led Outreach
  Interventions: Behavioral: Community Organization Led Outreach

INTERVENTIONS:
Behavioral: Healthcare Worker Focused Outreach — This a focused outreach intervention strategy specifically designed for healthcare workers.
  Other Names: Informational intervention
  Arms: Healthcare Worker Focused Outreach Intervention Strategy
Behavioral: Community Organization Led Outreach — This is a standard community engaged outreach approach that has traditionally been used in previous research. Analogous to the standard of care for outreach.
  Other Names: Informational intervention
  Arms: Community Organization Led Outreach

SUMMARY:
This mixed methods study evaluates the effectiveness and cost of a healthcare worker focused outreach intervention strategy versus community organization led outreach to explore contextual factors (individual, family, and community) affecting COVID-19 testing implementation outcomes and scalability.

DETAILED DESCRIPTION:
In Aim 2, the investigators conduct a mixed methods study to evaluate the effectiveness and cost of: (1) the healthcare worker focused outreach intervention strategy versus (2) community organization led outreach working with community based organizations. The investigators explore contextual factors (individual, family, and community) affecting COVID-19 testing implementation outcomes and scalability. The primary outcome is uptake of COVID-19 testing using the novel Rutgers Clinical Genomics Laboratory/RUCDR saliva test, the first FDA authorized diagnostic test using saliva to detect SARS-CoV-2 for non-invasive, home based self-testing. To compare participation rates in the two arms, our primary outcome, the investigators will use data on the number of tests performed per month up to a 12 month study period. For each intervention, the start time is the date of first attempted contact with potential participants and the end date is either the end of the study period, or the date at which the 1000th individual was tested (whichever comes first).

ELIGIBILITY:
Inclusion Criteria for Community Members and Healthcare Workers

* Self-identification as Black or Hispanic/Latino.
* Resident of Union, Passaic, Middlesex, or Essex County, NJ.
* Parent/legal guardian able to provide permission to participate for those under 18

Exclusion Criteria:

* Under 4 years of age.
* Unable to speak, understand, and/or read English or Spanish.
* Unable to provide informed consent/assent

Min Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2017 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Rutgers University, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jimenez ME, Rivera-Nunez Z, Crabtree BF, Hill D, Pellerano MB, Devance D, Macenat M, Lima D, Martinez Alcaraz E, Ferrante JM, Barrett ES, Blaser MJ, Panettieri RA Jr, Hudson SV. Black and Latinx Community Perspectives on COVID-19 Mitigation Behaviors, Testing, and Vaccines. JAMA Netw Open. 2021 Jul 1;4(7):e2117074. doi: 10.1001/jamanetworkopen.2021.17074. PMID 34264327
- [Background] Barrett ES, Andrews TR, Roy J, Greenberg P, Ferrante JM, Horton DB, Gordon M, Rivera-Nunez Z, Pellerano MB, Tallia AF, Budolfson M, Georgopoulos P, Reed D, Lynn B, Rosati R, Castaneda M, Dixon F, Pernell C, Hill D, Jimenez ME, Blaser MJ, Panettieri R Jr, Hudson SV. Community- Versus Health Care Organization-Based Approaches to Expanding At-Home COVID-19 Testing in Black and Latino Communities, New Jersey, 2021. Am J Public Health. 2022 Nov;112(S9):S918-S922. doi: 10.2105/AJPH.2022.306989. Epub 2022 Oct 20. PMID 36265092
- [Background] Rivera-Nunez Z, Jimenez ME, Crabtree BF, Hill D, Pellerano MB, Devance D, Macenat M, Lima D, Gordon M, Sullivan B, Rosati RJ, Ferrante JM, Barrett ES, Blaser MJ, Panettieri RA Jr, Hudson SV. Experiences of Black and Latinx health care workers in support roles during the COVID-19 pandemic: A qualitative study. PLoS One. 2022 Jan 18;17(1):e0262606. doi: 10.1371/journal.pone.0262606. eCollection 2022. PMID 35041702
- [Derived] Juarez R, Phankitnirundorn K, Ramirez A, Peres R, Maunakea AK, Okihiro M. Vaccine-Associated Shifts in SARS-CoV-2 Infectivity Among the Native Hawaiian and Other Pacific Islander Population in Hawaii. Am J Public Health. 2022 Nov;112(S9):S896-S899. doi: 10.2105/AJPH.2022.306973. Epub 2022 Sep 15. PMID 36108254

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From May through December 2021, 2017 eligible New Jersey residents registered for and consented to be part of an on-line study with a single questionnaire (including items on sociodemographic characteristics as well as COVID-19-related perceptions, behaviors, and challenges), after which they were able to order a free at-home saliva COVID-19 polymerase chain reaction test.
Pre-assignment Details: Some participants (n=917) chose not to participate in the questionnaire data collection and as a result were not assigned to a study arm after consent.
Period: Overall Study
Arm/Group | Healthcare Worker Focused Outreach Intervention Strategy | Community Organization Led Outreach
Started | 63 | 1037
Completed | 23 | 211
Not Completed | 40 | 826
Not completed — Lost to Follow-up | 40 | 826

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthcare Worker Focused Outreach Intervention Strategy | Community Organization Led Outreach | Total
Number analyzed (Participants) | 23 | 211 | 234
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 37 [18 to 51] | 44 [26 to 63] | 40.5 [22 to 57]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 157 | 173
  Male | 7 | 54 | 61
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black, non-Latino | 9 | 133 | 142
  Latino, non-Black | 11 | 65 | 76
  Black and Latino | 3 | 13 | 16

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Complete COVID-19 Testing
Description: Number of participants who return their saliva testing kit.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Healthcare Worker Focused Outreach Intervention Strategy | Community Organization Led Outreach
Number analyzed (Participants) | 63 | 1037
Participants | 23 | 211
Statistical Analysis 1: Comparison: Healthcare Worker Focused Outreach Intervention Strategy vs Community Organization Led Outreach; Test type: Superiority; p < 0.05, Regression, Logistic; Odds Ratio (OR) = 0.45, 95% CI 2-sided [0.17 to 1.23] — Healthcare Arm is the reference category

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Healthcare Worker Focused Outreach Intervention Strategy | Community Organization Led Outreach
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/211
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/211
Other Adverse Events (participants affected / at risk) | 0/23 | 0/211

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-21): https://cdn.clinicaltrials.gov/large-docs/33/NCT04766333/Prot_SAP_000.pdf